CLINICAL TRIAL: NCT01389882
Title: Application of Neurally Adjusted Ventilatory Assist (NAVA) in Preterm Infants and Assessment of Its Benefits Compared to Synchronized Intermittent Mandatory Ventilation (SIMV) With Pressure Support (PS)
Brief Title: Randomized Crossover Study of Neurally Adjusted Ventilatory Assist (NAVA) in Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Assist Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: VENT-01-NAVA
Record Dates: First submitted 2011-07-01; First posted 2011-07-08 (Estimated); Results first posted 2011-10-28 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Infant, Preterm
Keywords: mechanical ventilation; diaphragm electrical activity; pressure support
MeSH Terms: conditions — Premature Birth | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ventilator assist (Experimental)
  Interventions: Procedure: neurally adjusted ventilatory assist (NAVA) ventilator mode

INTERVENTIONS:
Procedure: neurally adjusted ventilatory assist (NAVA) ventilator mode — Neurally adjusted ventilatory assist (NAVA) utilizes the electrical activity of the diaphragm (EAdi) to trigger and cycle-off breaths, and therefore presents a means of bypassing the ventilator circuit, and the inherent delays with pneumatic triggering. This is a processed signal, which is not artificially influenced by changes in muscle length, chest wall configuration, and/or lung volume. It represents the summation of muscle motor unit recruitment and/or firing rate, and correlates with phrenic nerve activity. In this mode, the amount of support pressure is coupled with the magnitude of the EAdi. The proportion of support pressure to EAdi (NAVA level) is adjustable.
  Other Names: Servo-i (Maquet Critical Care AB, Solna, Sweden)

SUMMARY:
The purpose of this study is to test the hypothesis that neurally adjusted ventilatory assist (NAVA) will allow to lower the ventilator pressure at equivalent fractions of inspiratory oxygen (FiO2) and partial pressure of CO2 of capillary blood in preterm infants in comparison with currently used standard ventilation (synchronized intermittent mandatory ventilation with pressure-support ventilation, SIMV+PSV).

DETAILED DESCRIPTION:
The investigators will apply crossover comparison in preterm infants who received a ventilatory support. In patient whose frequency of mandatory support is under 25, the two ventilatory modes (SIMV+PSV and NAVA) are delivered by the same ventilator (Servo-I; Maquet Critical Care AB, Solna, Sweden) and will set to maintain similar blood gas analysis results.

Determination of the type of ventilatory mode used is performed using a cluster randomization. The randomized order of ventilatory mode will be used during total 9 hours; one mode for 4 hours and another mode for 5 hours. To rule out carry-over effects, a 1-hour interval for washout was guaranteed between modes. Recordings will be obtained over a total 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants mechanically ventilated
* ventilatory set frequency is under 25
* with informed consent of their parents

Exclusion Criteria:

* major congenital anomalies
* patients without self respiratory effort
* use of sedative or anesthetic drugs
* grade III or IV intraventricular hemorrhage
* phrenic nerve palsy or insufficiency

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Suk Kim, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a neonatal intensive care unit (NICU) of Seoul National University Hospital, in Seoul, Republic of Korea between March 2011 to July 2011.
Pre-assignment Details: 26 patients enrolled; 24 assigned to randomization and 2 excluded (1 extubated prior to the study and 1 developed exclusion criteria)
Groups:
- SN Group: Synchronized intermittent mandatory ventilation (SIMV) with Pressure support (PS) first, then Neurally adjusted ventilatory assist (NAVA)
- NS Group: NAVA first, then SIMV with PS
Period: Overall Study
Arm/Group | SN Group | NS Group
Started | 13 | 11
Completed | 12 | 7
Not Completed | 1 | 4
Not completed — Respiratory rate > 80/min during study | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SN Group | NS Group | Total
Number analyzed (Participants) | 13 | 11 | 24
Age Continuous [Median (Full Range); unit: days] | 7 [2 to 57] | 5 [2 to 70] | 5 [2 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 6 | 11 | 17
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 13 | 11 | 24
Gestational Age [Mean (Standard Deviation); unit: days] | 206 (28) | 212 (20) | 209 (24)
Birth Weight [Median (Full Range); unit: g] | 990 [370 to 2510] | 1630 [710 to 2510] | 1075 [370 to 2510]
Birth Height [Mean (Standard Deviation); unit: cm] | 37.2 (5.9) | 38.3 (6.7) | 37.7 (6.2)
Study Day Postmenstrual Age [Mean (Standard Deviation); unit: days] | 220 (20) | 222 (15) | 221 (18)
Study Day Body Weight [Median (Full Range); unit: g] | 1210 [670 to 2530] | 1530 [750 to 2580] | 1355 [670 to 2580]
Capillary Blood pH [Mean (Standard Deviation); unit: pH] | 7.31 (0.04) | 7.34 (0.06) | 7.32 (0.05)
Capillary Blood pCO2 [Mean (Standard Deviation); unit: mmHg] | 48.83 (8.93) | 44.45 (6.34) | 46.8 (8.00)
Capillary Blood pO2 [Mean (Standard Deviation); unit: mmHg] | 37.77 (7.03) | 37.00 (8.80) | 37.42 (7.72)
Capillary Blood HCO3 [Mean (Standard Deviation); unit: mmol/L] | 24.20 (3.45) | 21.62 (9.34) | 23.02 (6.78)

OUTCOME MEASURES:

1. Primary Outcome: Peak Inspiratory Pressure
Description: peak inspiratory pressure measured by a ventilator for 4 hours with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- SIMV With PS: synchronized intermittent mandatory ventilation with pressure support
- NAVA: neurally adjusted ventilatory assist
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
cmH2O | 13.45 (3.44) | 12.45 (2.66)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.043, Paired t-test; Mean Difference (Final Values) = 1.007, 95% CI 2-sided [0.036 to 1.978], Standard Deviation 2.015

2. Secondary Outcome: Mean Airway Pressure
Description: mean airway pressure measured by a ventilator for 4 hours with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
cmH2O | 7.99 (1.33) | 8.02 (1.23)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.245, Paired t-test; Median Difference (Final Values) = -0.232, 95% CI 2-sided [-0.637 to 0.174], Standard Deviation 0.841

3. Secondary Outcome: Minute Ventilation
Description: Minute ventilation measured by a ventilator for 4 hours with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: L/min/Kg
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
L/min/Kg | 0.53 (0.15) | 0.51 (0.11)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.257, Paired t-test; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.020 to 0.714], Standard Deviation 0.095

4. Secondary Outcome: Expiratory Tidal Volume
Description: Expiratory tidal volume measured by a ventilator for 4 hours with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: mL/Kg
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
mL/Kg | 8.73 (2.08) | 8.54 (2.24)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.601, Paired t-test; Mean Difference (Final Values) = 0.188, 95% CI 2-sided [-0.554 to 0.931], Standard Deviation 1.541

5. Secondary Outcome: Dynamic Compliance
Description: Dynamic Compliance measured by a ventilator for 4 hours with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
mL/cmH2O | 1.70 (0.47) | 1.84 (0.36)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.085, Paired t-test; Mean Difference (Final Values) = -0.149, 95% CI 2-sided [-0.320 to 0.023], Standard Deviation 0.355

6. Secondary Outcome: Work of Breathing
Description: Work of breathing of patients measured by a ventilator for 4 hours with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Median (Full Range); unit: mJ/L
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
mJ/L | 11.13 [3.92 to 60.79] | 8.38 [1.60 to 30.21]
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.002, Wilcoxon signed-rank test; Mean Difference (Final Values) = 6.516, 95% CI 2-sided [1.799 to 11.232], Standard Deviation 9.786

7. Secondary Outcome: Peak EAdi
Description: Peak electrical activity of the diaphragm
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
uV | 13.39 (5.68) | 11.70 (5.72)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.009, Paired t-test, 2-sided; Mean Difference (Final Values) = 1.69, 95% CI 2-sided [0.478 to 2.904], Standard Deviation 2.516

8. Secondary Outcome: Fraction of Oxygen
Description: Fraction of oxygen measured by a ventilator for 4 hours with each ventilator mode
Time Frame: four hours
Measure: Median (Full Range); unit: percentage of concentration
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
percentage of concentration | 23.33 [21.08 to 41.18] | 23.47 [20.75 to 39.07]
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.314, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.692, 95% CI 2-sided [-0.364 to 1.749], Standard Deviation 2.192

9. Secondary Outcome: Capillary Blood pH
Description: Capillary blood pH checked immediately after the 4-hour respiratory support with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
pH | 7.327 (0.051) | 7.334 (0.046)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.515, Paired t-test; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.030 to 0.016], Standard Deviation 0.047

10. Secondary Outcome: Capillary Blood pCO2
Description: Capillary blood pCO2 checked immediately after the 4-hour respiratory support with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
mmHg | 46.75 (7.43) | 46.64 (7.87)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.949, Paired t-test; Mean Difference (Final Values) = 0.1105, 95% CI 2-sided [-3.505 to 3.726], Standard Deviation 7.501

11. Secondary Outcome: Capillary Blood pO2
Description: Capillary blood pO2 checked immediately after the 4-hour respiratory support with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
mmHg | 38.89 (8.82) | 37.84 (8.51)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.709, Paired t-test; Mean Difference (Final Values) = 1.053, 95% CI 2-sided [-4.770 to 6.875], Standard Deviation 12.081

12. Secondary Outcome: Capillary Blood HCO3
Description: Capillary blood HCO3 checked immediately after the 4-hour respiratory support with each ventilator mode
Time Frame: four hours
Population: The analysis was "per protocol". 19 patients who had completed the study was used for the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | SIMV With PS | NAVA
Number analyzed (Participants) | 19 | 19
mmol/L | 24.46 (3.95) | 24.74 (3.57)
Statistical Analysis 1: Comparison: SIMV With PS vs NAVA; Test type: Superiority or Other; p = 0.600, Paired t-test; Mean Difference (Final Values) = -0.274, 95% CI 2-sided [-1.350 to 0.802], Standard Deviation 2.233

ADVERSE EVENTS:
Arm/Group | SN Group | NS Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

LIMITATIONS AND CAVEATS:
Two patients were excluded prior to the study and five patients were interrupted the study because of a developed exclusion criterion during the protocol. Because of eliminated participants, the number of subjects analyzed was reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No